CLINICAL TRIAL: NCT04930250
Title: A Randomised, Double-blind, Controlled, Crossover Study to Evaluate the Acute Effect on Glycemic Response and Related Biomarkers When Replacing Rapidly Digested Carbohydrates by β-glucan-rich Oat Bran Processed in Different Conditions
Brief Title: Effect of Various Processed Oat Bran in a Beverage Matrix on Glycaemic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: National University Hospital, Singapore (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20.13.DAI
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomised controlled, double-blind, full crossover study conducted in an acute setting. 20 subjects will receive 5 test products, over 5 separate test visits in a crossover design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The test products are coded by group coding (A - E).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Oat bran fibre processed with method A (Experimental): Beverage powder with 12% oat bran processed with method A
  Interventions: Other: Beverage powder with 12% oat bran processed with method A
- Oat bran fibre processed with method B (Experimental): Beverage powder with 12% oat bran processed with method B
  Interventions: Other: Beverage powder with 12% oat bran processed with method B
- Oat bran fibre processed with method C (Experimental): Beverage powder with 12% oat bran processed with method C
  Interventions: Other: Beverage powder with 12% oat bran processed with method C
- Minimally-processed oat bran (positive control) (Active Comparator): Beverage powder with minimally-processed oat bran (Positive Control)
  Interventions: Other: Placebo Comparator: Minimally-processed oat bran (Positive Control)
- Readily-digestible carbohydrate (negative control) (Placebo Comparator): Beverage powder with readily digestible carbohydrate (Negative Control)
  Interventions: Other: Placebo Comparator: Readily-digestible carbohydrate (negative control)

INTERVENTIONS:
Other: Beverage powder with 12% oat bran processed with method A — 50g of beverage powder to be reconstituted with 330ml of water. Subjects will orally consume one of the five test products in a random order over the five test visits.
  Arms: Oat bran fibre processed with method A
Other: Beverage powder with 12% oat bran processed with method B — 50g of beverage powder to be reconstituted with 330ml of water. Subjects will orally consume one of the five test products in a random order over the five test visits.
  Arms: Oat bran fibre processed with method B
Other: Beverage powder with 12% oat bran processed with method C — 50g of beverage powder to be reconstituted with 330ml of water. Subjects will orally consume one of the five test products in a random order over the five test visits.
  Arms: Oat bran fibre processed with method C
Other: Placebo Comparator: Minimally-processed oat bran (Positive Control) — 50g of beverage powder to be reconstituted with 330ml of water. Subjects will orally consume one of the five test products in a random order over the five test visits.
  Arms: Minimally-processed oat bran (positive control)
Other: Placebo Comparator: Readily-digestible carbohydrate (negative control) — 50g of beverage powder to be reconstituted with 330ml of water. Subjects will orally consume one of the five test products in a random order over the five test visits.
  Arms: Readily-digestible carbohydrate (negative control)

SUMMARY:
Whilst a cause-and-effect relationship between consumption of oat ß-glucans and reduction in PPGR has been demonstrated, little is understood about its:

* Application to liquid matrices: There are few studies which looked into the effect of a dose of ß-glucan applicable to beverages. Previous studies have explored oat ß-glucan doses between 2g to 13g per serving of test product (Note: the oat ß-glucan dose for the proposed trial is <2g).
* Impact following processing: Collectively, oat processing, ß-glucan structure and its physiological impact on PPGR are closely linked. Some studies have investigated the effect of oat processing or dosage on PPGR, but to our knowledge, no study has systematically characterised the effect of processing on oat structure, and clinically measured its subsequent impact on PPGR.

DETAILED DESCRIPTION:
The proposed study is a randomised, double blind, controlled, crossover trial to investigate the postprandial effects on glycemic response and related biomarkers/biological surrogates in five test product beverages:

This study will investigate the post-prandial effects of five test products, including two controls:

1. Beverage powder with 12% oat bran processed with method A (Test Product: TP-1)
2. Beverage powder with 12% oat bran processed with method B (Test Product: TP-2)
3. Beverage powder with 12% oat bran processed with method C (Test Product: TP-3)
4. Beverage powder with 12% minimally-processed oat bran (Positive Control) (Test Product: TP-PC)
5. Beverage powder without oat bran (Negative Control) (Test Product: TP-NC)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, age between 24 and 39 years
2. Healthy individuals with no comorbidities or on regular medication
3. BMI between 18.5-25 kg/m2
4. Able to understand and willing to sign an informed consent form in English
5. Regularly consume breakfast
6. Able and willing to consume 330ml of liquid in 10 minutes
7. For female participants, have a regular menstrual cycle

Exclusion Criteria:

1. Known food allergies or intolerances specifically to gluten, milk, lactose or any grains
2. Known drug allergies specifically paracetamol
3. Known sensitivity or has had an adverse reaction to paracetamol and non-steroidal anti-inflammatory drugs (NSAID) in the past
4. Individuals with regular prescriptions or regularly consume medication (at least once a month), including alternative medicine (e.g. traditional Chinese medicine)
5. Had been diagnosed or with a history of any metabolic disease or disorders, including diabetes, gestational diabetes and hypertension
6. Had been diagnosed or with a history of gastrointestinal disorders e.g. irritable bowel syndrome, constipation, diverticulitis
7. Had been hospitalised in the 3 months prior to the study.
8. Pregnant or lactating women, or planning to conceive in the next 3 months
9. Consumes more than 2 alcoholic drinks per day i.e. one drink is defined as either 150ml of wine, 340ml of beer/cider or 45ml of distilled spirit.
10. Smokers
11. Poor peripheral venous access based on past experiences with blood draw
12. Significant change in weight (≥ 3 kg body weight) in the past 3 months
13. Significant exercise pattern over the past 3 months defined as high-intensity exercise of more than 3 hours per week
14. Currently on a specialised diet e.g. vegetarian, vegan, weight loss plan, high protein diet
15. Unwilling to refrain from consuming fibre or prebiotic supplements, high fibre ingredients and more than 5 servings of fruits and vegetables per day over the length of the study.
16. Has donated blood in the past one month
17. Hierarchical link with the research team members
18. Participating in another clinical study

Ages: 24 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response - Area under the plasma concentration versus time curve (AUC) | through study completion, an average of 7 months
  Postprandial glycemic response reflected by 3-hour area under the plasma concentration versus time curve (AUC) assessed over all cross-sectional blood glucose values (i.e. T0/T15/T30/T45/T60/T90/T120/T180).
Postprandial glycemic response - Peak Plasma Concentration (Cmax) | through study completion, an average of 7 months
  Postprandial glycemic response by the peak plasma concentration (Cmax) assessed over a 3-hour period by all cross-sectional blood glucose values (i.e. T0/T15/T30/T45/T60/T90/T120/T180).
Postprandial glycemic response - Time to Peak Plasma Concentration (Tmax) | through study completion, an average of 7 months
  Postprandial glycemic response reflected by time to achieve the peak plasma concentration (Tmax) assessed over a 3-hour period by all cross-sectional blood glucose values (i.e. T0/T15/T30/T45/T60/T90/T120/T180).

SECONDARY OUTCOMES:
Postprandial insulin response (PPIR) | through study completion, an average of 7 months
  PPIR over a 3-hour period
Postprandial blood gastric inhibitory polypeptide (GIP) | through study completion, an average of 7 months
  Postprandial blood GIP over a 3-hour period
Postprandial blood glucagon-like peptide 1 (GLP-1) | through study completion, an average of 7 months
  Postprandial blood GLP-1 over a 3-hour period
Gastric emptying rate | through study completion, an average of 7 months
  Gastric emptying rate measured through postprandial blood paracetamol concentration over a 4-hour period
Satiety | through study completion, an average of 7 months
  Satiety assessed via a Visual Analogue Scale questionnaire from 0-10 over a 4-hour period, with 0 being least satiated and 10 being most satiated
Gastrointestinal comfort | through study completion, an average of 7 months
  Gastrointestinal comfort assessed via a Visual Analogue Scale questionnaire from 0-10 over a 4-hour period, with 0 being lowest discomfort and 10 being greatest discomfort
Ingredient fermentability by colonic bacteria | through study completion, an average of 7 months
  Fermentability by colonic bacteria will be assessed via breath hydrogen and methane (ppm) levels over a 4-hour period

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided